CLINICAL TRIAL: NCT00131807
Title: A Study to Explore the Association Between Blood Pressure, HIV and Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: The Hypertension Trust (Unknown)
Other Study IDs: NPSW03
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2007-04

CONDITIONS: HIV Infections
Keywords: Blood Pressure; HIV; Antiretroviral therapy
MeSH Terms: conditions — HIV Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Blood Pressure Measurement
Procedure: Questionnaire

SUMMARY:
The purpose of this study is to explore the association between blood pressure, HIV and/or its treatment in a cross sectional observational study.

DETAILED DESCRIPTION:
Deaths from AIDS have declined dramatically since the introduction of highly active antiretroviral therapy in HIV infected patients. However the incidence of heart disease has increased four-fold and is now one of the major causes of death in HIV infected patients. While HIV drugs are known to adversely affect serum lipids, the evidence concerning the association between raised blood pressure (a major risk for cardiovascular disease) HIV and/or its treatment is limited and conflicting. The researchers believe it of interest to study heart disease risk factors in patients with HIV infection to avoid one premature cause of death (AIDS) being replaced with another potentially preventable cause of death and disability (heart disease). In this cross sectional observational study the researchers will systematically measure blood pressure and other cardiovascular risk factors in HIV positive patients on and off antiretroviral therapy. These individuals will be matched for age, sex and ethnic group with HIV negative individuals.

ELIGIBILITY:
Inclusion Criteria:

* Attending St. Mary's sexual health outpatient department
* Patients willing to give written informed consent
* Ability to communicate in English

Exclusion Criteria:

* Failure to give written informed consent in English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000
Dates: Start 2005-09; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil R Poulter, Principal Investigator — Imperial College London
Locations (1):
- St. Mary's Hospital, Paddington, London, United Kingdom